CLINICAL TRIAL: NCT05107011
Title: A Multicenter, Open-label, Phase I/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of LBL-015 in Patients With Advanced Malignant Tumors.
Brief Title: Phase I/II Clinical Trial of LBL-015 for Injection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nanjing Leads Biolabs Co.,Ltd (Industry)
Collaborators: Shanghai East Hospital (Other); Shandong Cancer Hospital and Institute (Other); Henan Cancer Hospital (Other Government); Hunan Cancer Hospital (Other); The First Affiliated Hospital of Nanchang University (Other); The First Affiliated Hospital of Bengbu Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LBL-015-CN-001
Record Dates: First submitted 2021-10-20; First posted 2021-11-04 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Advanced Malignant Tumor
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LBL-015 (Experimental): Drug: LBL-015 for Injection，Initial dose - MTD; Q2W
  Interventions: Drug: LBL-015 for Injections

INTERVENTIONS:
Drug: LBL-015 for Injections — Initial dose - MTD ; Q2W ; intravenous infusion
  Other Names: LBL-015

SUMMARY:
A Multicenter, Open-label, Phase I/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of LBL-015 in Patients With Advanced Malignant Tumors.

DETAILED DESCRIPTION:
This study is a single-arm, open-label, multi-center, dose-escalation and expansion phase I/II study to evaluate the safety, tolerability, pharmacokinetic characteristics, receptor occupancy, immunogenicity and efficacy of LBL-015 in patients with advanced malignant tumors.About 202 patients with advanced malignant tumor will be enrolled.

The study is divided into Phase I study stage (dose escalation/PK expansion stage) and Phase II study stage (indication expansion stage).

Patients with advanced or metastatic advanced malignant tumor who have failed previous standard treatment, are not suitable for standard treatment or have no standard treatment are included in the phase I study.

After obtaining the RP2D in Phase I study ,Phase II study stage (indication expansion stage) was initiated.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to follow the trial treatment regimen and visit schedule, voluntarily enroll in the study, and sign the written informed consent form；
2. Age ≥18 and ≤75 years old at the time of signing the informed consent form, regardless of gender;
3. Have a performance status of 0 to 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status Scale；
4. Have a life expectancy of at least 12 weeks；
5. There is adequate organ and bone marrow function,Conforms to laboratory test results;
6. Fertile men and women of childbearing age are willing to take effective contraceptive measures (including abstinence, intrauterine devices, hormonal contraception, and correct use of condoms) from the signing of the informed consent form to 6 months after the last dose of the investigational drug; women of childbearing age include premenopausal women and women who had menopause less than two years ago. Blood pregnancy test results must be negative for women of childbearing age within 7 days prior to the initial dose of the investigational drug.

Exclusion Criteria:

1. Received other unapproved investigational drug or treatment within 4 weeks prior to first dose of investigational drug；
2. Subjects who underwent major organ surgery (excluding needle biopsy) or significant trauma within 4 weeks prior to the initial use of the investigational drug, or require elective surgery during the trial period；
3. Use of immunomodulatory drugs within 14 days prior to the initial use of the investigational drug, including but not limited to thymosin, interleukin, and interferon；
4. Subjects with an active infection that currently requires intravenous anti infective therapy；
5. History of immunodeficiency, including positive HIV antibody test results；
6. Pregnant or lactating women；
7. The investigator's assessment that there may be other factors affecting compliance among participants or that some may not be suitable for inclusion in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 28 days after the first dose.
  MTD is defined as the hightest dose level at which no more than 1 out of 6 subjects experiences a DLT during the first cycles. It was used to evaluate the tolerability.
Dose-limiting toxicities（DLT） | 28 days after the first dose
  DLT describes side effects of a drug or other treatment that are serious enough to prevent an increase in dose or level of that treatment. It was used to evaluate the safety.

SECONDARY OUTCOMES:
Cmax | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (30 days after drug withdrawal or before the start of new anti-tumor therapy
  Maximum serum concentration
Tmax | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (30 days after drug withdrawal or before the start of new anti-tumor therapy
  After taking a single dose, Time to reach maximum plasma concentration
immunogenicity | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (30 days after drug withdrawal or before the start of new anti-tumor therapy
  The immunogenicity is evaluated by the incidence of anti-drug antibodies (ADA) and neutralizing antibodies (if applicable) in subjects.
Pharmacodynamic (PD) index | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (30 days after drug withdrawal or before the start of new anti-tumor therapy
  Evaluate the receptor occupancy of the drug

CONTACTS AND LOCATIONS:
Overall Officials: Jin li, Principal Investigator — Shanghai East Hospital
Locations (6):
- China (6):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shanghai East Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No